CLINICAL TRIAL: NCT05325840
Title: Evaluation of the Effect of Music Played During the Non-Stress Test on Fetal Health, Anxiety Level of the Pregnant and Blood Pressure
Brief Title: Non Stress Test and Music Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Sibel ÖZTÜRK, Asst. Prof., Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Ataturk University SÖZTÜRK0002
Record Dates: First submitted 2022-01-31; First posted 2022-04-13 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Fetal Health; Pregnancy Related
Keywords: music; pregnancy; nonstrest test; fetal; health

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music therapy (Experimental): Experimental Group: Pre-test will be applied to pregnant women before the intervention. Since ST will be applied later, Nki will be applied to pregnant women, and their props will then be right lateral or lateral. NST registration form will be filled.
  After the pregnancy is given, the type of music (Classical Turkish Music, Turkish Classical Music, Lullaby) is asked according to the preferences of the pregnant women and their music is given for 20 minutes. The NST process will be implemented from start to finish. In the application, music from pregnant women will be played on MP3 players. After the NST procedure is applied, the pregnant women will have a son.
  Interventions: Other: music terapy
- standard of care (No Intervention): Control group: First of all, Personal Information Form, State Anxiety Scale and blood pressure measurement will be made to the pregnant women in the control group. In order to perform the NST procedure, the pregnant women will be given the left side or right side position to fix the probes. NST registration form will be filled.
  20 minutes after positioning the pregnant women. During the routine NST procedure will be applied and no intervention will be made. After the NST procedure is completed, the State Anxiety Scale and blood pressure measurement will be repeated as the last test of the pregnant women.

INTERVENTIONS:
Other: music terapy — The aim of this study was to examine the effects of the music concert applied during the nonstress test procedure on the health of the fetus, the anxiety level of the pregnant woman and blood pressure.
  Arms: music therapy

SUMMARY:
Today, many methods are used in the evaluation of intrauterine fetal well-being. Non-stress test (NST) method is mostly used in the non-invasive evaluation of fetal well-being during pregnancy and labor. NST is a procedure in which fetal heart sounds are recorded and the relationship between fetal movements and fetal heart beat is monitored.3 Various methods are used to minimize the psychological effects that occur during pregnancy. Among these methods, it has been seen in the studies in the literature that music, which is a non-pharmacological method, has a positive effect on the pregnant woman and the fetus. It is easy and enjoyable to listen to music during the routine non-stress test process. However, there are not enough studies to prove the effect of music.

The aim of this study was to examine the effects of the music concert applied during the nonstress test procedure on the health of the fetus, the anxiety level of the pregnant woman and blood pressure.

DETAILED DESCRIPTION:
expected

ELIGIBILITY:
Inclusion Criteria:

* Become literate
* Be in the 18-45 age range.
* Being at the 32nd and above gestational week
* Not carrying any risk factors during pregnancy (preeclampsia, IUGR, gestational diabetes, etc.)
* Have eaten at least two hours before the NST procedure
* No fetal defined cardiovascular disease
* The pregnant woman is open to communication and does not have mental or mental problems.
* Absence of auditory problems

Exclusion Criteria:

* Absence of illiteracy of the pregnant woman
* Uterine contraction in NST
* Pregnant women who need fetal distress and urgent intervention by the physician

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — woman
Enrollment: 140 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Effect of Music Played During the Non-Stress Test on Fetal Health, Anxiety Level of the Pregnant and Blood Pressure | Day 1
  The research is an experimentally planned randomized controlled trial.The sample of the study consists of pregnant women (69 experimental group, 68 control group) between 32nd and 41st weeks. The pregnant women were evaluated with the state anxiety scale. The scale consists of 20 items in total. Scoring is calculated by subtracting the total weighted score for the reverse statements from the total weighted score for the direct statements. A predetermined invariant value is added to this obtained number.This value is 50 for the state anxiety scale. The most recent value is the individual's anxiety score. As the score obtained from the scale increases, it indicates that the level of anxiety increases. 0-19 point no anxiety, 20-39 points mild anxiety, 40-59 points moderate anxiety, 60-79 points severe anxiety, 80 points severe anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Bingöl Solhan Devlet Hastanesi, Bingöl, Solhan Bingöl, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No